CLINICAL TRIAL: NCT00439608
Title: Cetuximab, Paclitaxel, Carboplatin and Radiation for Esophageal, Gastroesophageal Junction and Gastric Cancer BMS#CA225091
Brief Title: Cetuximab, Paclitaxel, Carboplatin & Radiation for Esoph, Gastroesoph & Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, howard safran, Principal Investigator, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-EG-203; BMS#CA225091 (Other: BMS); NCT01904435 (obsolete NCT alias)
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: esophageal cancer; gastroesophageal cancer; gastric cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Cetuximab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Cetuximab, paclitaxel, and carboplatin weekly for 6 weeks with 50.4 Gy radiation.
  Interventions: Drug: Cetuximab,Paclitaxel, Carboplatin

INTERVENTIONS:
Drug: Cetuximab,Paclitaxel, Carboplatin — IV treatment for 6 weeks

SUMMARY:
Cetuximab, Paclitaxel, Carboplatin and Radiation for Esophageal, Gastroesophageal Junction and Gastric Cancer

DETAILED DESCRIPTION:
The primary objective of this phase II trial is to estimate the rate of complete pathologic response as determined by surgical resection or post treatment endoscopy (for patients not undergoing resection) for the treatment regimen being tested. With a total accrual of 28 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients are required to have pathologically confirmed adenocarcinoma or squamous cell carcinoma of the esophagus, gastroesophageal junction, or stomach.
* Patients may have mediastinal, celiac adenopathy, peri-portal and regional gastric lymphadenopathy.
* There must be no evidence of distant organ metastases.
* No prior radiation for gastric or esophageal cancer.
* Patients must be > 18 years of age, and nonpregnant
* Patients must have an ANC > 1,500/ul, platelets > 100,000/ul, creatinine < 2 x upper limit normal (ULN) and bilirubin < 1.5 x ULN, and AST < 3 x ULN.
* ECOG performance status 0-2.
* Patients must not have significant infection or other coexistent medical condition that would preclude protocol therapy.
* Female patients, must either be not of child bearing potential or have a negative pregnancy test within 7 days of starting study treatment. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal. Pregnant or lactating females are not eligible.
* All patients must sign informed consent

Exclusion Criteria:

Any of the following criteria will make the patient ineligible to participate in this study:

* Acute hepatitis or AIDS.
* Active or uncontrolled infection.
* Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
* Prior therapy which specifically and directly targets the EGFR pathway.
* Prior severe infusion reaction to a monoclonal antibody.
* Any concurrent chemotherapy not indicated in the study protocol or any other investigational agent(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — Brown University
Locations (1):
- Brown University Oncology Group, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 patients were enrolled at multiple hospitals and medical clinics
Groups:
- Treatment: Cetuximab, Paclitaxel, Carboplatin and Radiation for Esophageal, Gastroesophageal Junction and Gastric Cancer
  Patients received cetuximab, 400 mg/mg2 over 2 h on Day 1 then 250 mg/m2/week over 1 h, for 5 additional weeks. Patients also received paclitaxel, 50 mg/m2/week, over 1 h and carboplatin AUC (area under the curve) = 2/week, over 30 min, for 6 weeks. Cetuximab was administered first. Patients were then monitored for 1 h. Paclitaxel was then administered followed by carboplatin. Radiation was generally administered after chemotherapy. Dexamethasone 20 mg intravenously (IV), diphenhydramine 50 mg IV, and ranitidine 50 mg IV were given 30 min before treatment. Dosages of dexamethasone and diphenhydramine could be reduced in subsequent weeks if no hypersensitivity reactions were observed.
Period: Overall Study
Arm/Group | Treatment
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients received cetuximab, 400 mg/mg2 over 2 h on Day 1 then 250 mg/m2/week over 1 h, for 5 additional weeks. Patients also received paclitaxel, 50 mg/m2/week, over 1 h and carboplatin AUC (area under the curve) = 2/week, over 30 min, for 6 weeks. Cetuximab was administered first.
Arm/Group | Treatment
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 50
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Reponse Rate at Time of Surgery by Tissue
Description: pathologic complete response rate at surgery
Time Frame: within 30 days of last treatment
Measure: Number; unit: participants
Groups:
- Treatment: Cetuximab, Paclitaxel, Carboplatin and Radiation for Esophageal, Gastroesophageal Junction and Gastric Cancer
Arm/Group | Treatment
Number analyzed (Participants) | 57
participants | 40

2. Secondary Outcome: Number of Participants With Grade 2 and/or 3 Rash in Patients With Adenocarcinoma or Squamous Cell Carcinoma of the Esophagus, Gastroesophageal Junction, or Stomach.
Description: CTCAE version 3: grade 2 and 3 rash. This is reported as it was the most common toxicity.
Time Frame: baseline, then during treatment, about 5 weeks through 30 days post treatment.
Population: 60 patients were analyzed for toxicity but 57 for overall response.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 60
participants | 37

ADVERSE EVENTS:
Time Frame: For 30 days post end of treatment, approximately 6 months.
Description: CTCAE v 3
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 2/60
Serious Adverse Events (participants affected / at risk) | 7/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=60)
esophagitis (Gastrointestinal disorders) | 1 (1) — grade 4 esophagitis
ANC (Blood and lymphatic system disorders) | 2 (2)
anemia (Blood and lymphatic system disorders) | 1 (1)
hypersensitivity cetuximab (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=60)
Rash (Skin and subcutaneous tissue disorders) | 37 (37) — This event is being reported as it is the most common toxicity > or = grade 2 that was reported in the manuscript.
esophagitis (Gastrointestinal disorders) | 30 (30)
dehydration (General disorders) | 29 (29)
fatigue (General disorders) | 21 (21)
anorexia (Metabolism and nutrition disorders) | 15 (15)
weight loss (Metabolism and nutrition disorders) | 10 (10)
nausea (General disorders) | 9 (9)
vomiting (General disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 3 (3)
constipation (Gastrointestinal disorders) | 5 (5)
Hypersensitivity (Investigations) | 9 (9) — To both paclitaxel and cetuximab
infection (Infections and infestations) | 7 (7)
fever (General disorders) | 3 (3)
hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 29 (29)
Thromobocytopenia (Blood and lymphatic system disorders) | 3 (3)
anemia (Blood and lymphatic system disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2006-04-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT00439608/Prot_SAP_ICF_000.pdf